CLINICAL TRIAL: NCT04605991
Title: A Study of LY900014 in Participants With Type 2 Diabetes Using Continuous Glucose Monitoring
Brief Title: A Study of Mealtime Insulin LY900014 in Participants With Type 2 Diabetes Using Continuous Glucose Monitoring (PRONTO-Time in Range)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17428; I8B-MC-ITSW (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY900014 (Experimental): LY900014 (100 units/milliliter (U/mL)) is a mealtime insulin administered subcutaneously (SC) 0-2 minutes prior to each meal in combination with insulin glargine (100 U/mL) SC as long-acting insulin. Mealtime (bolus) and long-acting (basal) insulin doses were titrated to achieve glucose targets during the study.
  Interventions: Drug: LY900014; Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY900014 — Administered SC
Drug: Insulin Glargine — Administered SC

SUMMARY:
This study is being done to evaluate glycemic control in participants with type 2 diabetes who are taking mealtime insulin LY900014 in combination with long-acting insulin glargine. Participants will use continuous glucose monitoring (CGM) (Freestyle Libre 14-day system) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed (clinically) with type 2 diabetes mellitus (T2D) for at least 1 year prior to screening.
* Have been treated with basal-bolus multiple daily injection (MDI) therapy for at least 90 days prior to screening including:

  * Basal insulin glargine U-100, in combination with bolus insulin analog (insulin lispro, insulin aspart, or insulin glulisine) with meals.
  * Participant must have been treated with the same type of allowed bolus insulin analog for at least 30 days prior to screening.
* Participants may be treated with up to 3 of the following oral antihyperglycemic medications (OAMs) for T2D in accordance with local regulations:

  1. Metformin
  2. Dipeptidyl peptidase-4 (DPP-4) inhibitor
  3. sodium glucose cotransporter 2 (SGLT2) inhibitor
  4. oral glucagon-like peptide 1 (GLP-1) agonist
* Doses of OAMs are required to have been stable for at least 90 days prior to screening.
* Participants may be treated with injectable GLP-1 receptor agonist for T2D in accordance with local regulations. The GLP-1 receptor agonist dose is required to have been stable for at least 90 days prior to screening.
* Have an HbA1c value ≥7.5% and ≤10% according to the central laboratory at screening.

Exclusion Criteria:

* Have been diagnosed at any time with type 1 diabetes mellitus or latent autoimmune diabetes in adults.
* Have had any episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within 6 months prior to screening.
* Have had any episode of hyperglycemic hyperosmolar state or diabetic ketoacidosis within 6 months prior to screening.
* Have hypoglycemia unawareness as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (29):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - AMCR Institute, Escondido, California
  - Valley Endocrine, Fresno, Fresno, California
  - University Clinical Investigators, Inc., Tustin, California
  - Coastal Metabolic Research Centre, Ventura, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - Encore Medical Research, Hollywood, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research at The Jones Center, Macon, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Research NYC, Inc, New York, New York
  - Suny Health Science Center at Syracuse, Syracuse, New York
  - Cataret Medical Group, Morehead City, North Carolina
  - Intend Research, LLC, Norman, Oklahoma
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Burke Internal Medicine and Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Manati Center for Clinical Research Inc, Manatí, PR
  - Advanced Clinical Research, LLC, Bayamón

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Bailey TS, Bode BW, Wang Q, Knights AW, Chang AM. Increased Time in Range with Ultra Rapid Lispro Treatment in Participants with Type 2 Diabetes: PRONTO-Time in Range. Diabetes Ther. 2023 May;14(5):883-897. doi: 10.1007/s13300-023-01400-w. Epub 2023 Apr 7. PMID 37029268
- See also: A Study of Mealtime Insulin LY900014 in Participants with Type 2 Diabetes Using Continuous Glucose Monitoring (PRONTO-Time in Range) — https://trials.lillytrialguide.com/en-US/trial/1o3M94i5GGiiJPY7Q2RZBo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY900014
Started | 187
Received at Least 1 Dose of Study Drug | 176
Completed | 154
Not Completed | 33
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 14
Not completed — Non-compliance with study | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY900014: LY900014 (100 U/mL) is a mealtime insulin administered SC 0-2 minutes prior to each meal in combination with insulin glargine (100 U/mL) SC as long-acting insulin. Mealtime (bolus) and long-acting (basal) insulin doses were titrated to achieve glucose targets during the study.
Arm/Group | LY900014
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 140
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 187
Percentage of Time With Sensor Glucose Values Between 70 and 180 mg/dL During Daytime Period [Mean (Standard Deviation); unit: Percentage of time] — Percentage of Time with Continuous Glucose Monitoring (CGM) Sensor Glucose Values between 70-180 mg/dL (3.9-10.0 millimoles/liter [mmol/L]) (both inclusive) during Daytime Period Population: All participants who received at least one dose of study drug and had baseline CGM glucose values.
  Percentage of time
    number analyzed (Participants) | 163
    (all) | 58.65 (15.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Time With Continuous Glucose Monitoring (CGM) Sensor Glucose Values Between 70-180 Milligrams/Deciliter (mg/dL) (3.9-10.0 Millimoles/Liter [mmol/L]) (Both Inclusive) During Daytime Period at Week 12
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline CGM glucose values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | LY900014
Number analyzed (Participants) | 153
Percentage of time | 3.8 (1.38)

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline HbA1c values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY900014
Number analyzed (Participants) | 167
Percentage of HbA1c | -0.44 (0.069)

3. Secondary Outcome: Change From Baseline in Percentage of Time With CGM Sensor Glucose Values Between 70-180 mg/dL (3.9-10.0 mmol/L) (Both Inclusive) During the 24-hour Period at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline CGM glucose values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | LY900014
Number analyzed (Participants) | 153
Percentage of time | 3.3 (1.37)

4. Secondary Outcome: Change From Baseline in Percentage of Time With CGM Sensor Glucose Values <54 mg/dL (<3.0 mmol/L) During Daytime and 24-hour Periods at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline CGM glucose values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | LY900014
Number analyzed (Participants) | 153
Percentage of time
  Daytime | 0.10 (0.117)
  24-hour Period | 0.00 (0.153)

5. Secondary Outcome: Change From Baseline in Percentage of Time With CGM Sensor Glucose Values >180 mg/dL (>10.0 mmol/L) During Daytime and 24-hour Period at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline CGM glucose values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | LY900014
Number analyzed (Participants) | 153
Percentage of time
  Daytime | -4.3 (1.49)
  24-Hour Period | -3.4 (1.51)

6. Secondary Outcome: Change From Baseline in Percentage of Time With CGM Sensor Glucose Value >250 mg/dL (>13.9 mmol/L) During Daytime and 24-hour Period at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline CGM glucose values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | LY900014
Number analyzed (Participants) | 153
Percentage of time
  Daytime | -1.56 (0.773)
  24-Hour Period | -1.07 (0.748)

7. Secondary Outcome: Change From Baseline in Postprandial Incremental Area Under the Glucose Curve (iAUC) 0-1 Hour at Week 12
Description: iAUC reflects the metabolic control and is calculated using the standard trapezoidal rule from Glucose measures taken every 15 minutes from 0 to 1 hour after meal using CGM sensor (i.e., 0, 15, 30, 45, 60 minutes after meal). LS mean was determined by ANCOVA (analysis of covariance) with Baseline as covariate.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline iAUC data.
Measure: Least Squares Mean (Standard Error); unit: milligrams*hours per deciliter (mg*h/dl)
Arm/Group | LY900014
Number analyzed (Participants) | 111
milligrams*hours per deciliter (mg*h/dl)
  Breakfast: number analyzed (Participants) | 107
  Breakfast | -1.57 (1.191)
  Lunch: number analyzed (Participants) | 108
  Lunch | -0.56 (1.205)
  Dinner: number analyzed (Participants) | 105
  Dinner | -2.76 (1.287)
  Overall - across meals | -2.46 (0.856)

8. Secondary Outcome: Change From Baseline in Postprandial Incremental Area Under the Glucose Curve (iAUC) 0-2 Hour at Week 12
Description: iAUC reflects the metabolic control and is calculated using the standard trapezoidal rule from glucose measures taken every 15 minutes from 0 to 2 hours after meal using CGM sensor (i.e., 0, 15, 30, 45, 60, 75, 90, 105, 120 minutes after meal). LS mean was determined by ANCOVA (analysis of covariance) with Baseline as covariate.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline iAUC data.
Measure: Least Squares Mean (Standard Error); unit: mg*h/dl
Arm/Group | LY900014
Number analyzed (Participants) | 111
mg*h/dl
  Breakfast: number analyzed (Participants) | 107
  Breakfast | -8.1 (3.78)
  Lunch: number analyzed (Participants) | 108
  Lunch | -2.57 (3.652)
  Dinner: number analyzed (Participants) | 104
  Dinner | -8.32 (3.933)
  Overall - across meals | -8.8 (2.47)

9. Secondary Outcome: Percentage of Participants With HbA1c <7% and ≤6.5%
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 12
Population: All participants who received at least one dose of study drug and had post-baseline HbA1c values.
Measure: Number; unit: Percentage of participants
Arm/Group | LY900014
Number analyzed (Participants) | 154
Percentage of participants
  HbA1c <7% | 16.88
  HbA1c ≤6.5% | 4.55

10. Secondary Outcome: Change From Baseline in Daily Insulin Dose at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: Units per day
Arm/Group | LY900014
Number analyzed (Participants) | 155
Units per day
  Basal Insulin Dose | 3.7 (1.29)
  Bolus Insulin Dose | 18.0 (2.53)
  Total Insulin Dose | 22.0 (3.26)

11. Secondary Outcome: Change From Baseline in Bolus/Total Insulin Dose Percentage at Week 12
Description: LS mean was determined by MMRM model with Baseline + Time as variables.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline values for bolus and total insulin dose.
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin dose
Arm/Group | LY900014
Number analyzed (Participants) | 154
percentage of insulin dose | 6.0 (0.97)

12. Secondary Outcome: Change From Baseline in Insulin Treatment Satisfaction Questionnaire (ITSQ) - Glycemic Control Domain Score at Week 12
Description: The ITSQ is a 22-item questionnaire that assesses treatment satisfaction for subjects taking insulin under 5 domains: Inconvenience of Regimen [IR - 5 items], Lifestyle Flexibility [LF - 3 items], Glycemic Control [GC - 3 items], Hypoglycemic Control [HC - 5 items], Insulin Delivery Device [IDD - 6 items]. Each Item is measured on a 7-point scale, with scores ranging for IR from 5 to 35, LF from 3 to 21, GC from 3 to 21, HC from 5 to 35, IDD from 6 to 42. Lower scores reflect better outcomes. Data presented are for Glycemic Control Domain Scores transformed on a 0-100 scale, where transformed domain score = 100×[(7-raw domain score)/6]. Higher scores indicate better glycemic control. Least squares (LS) mean estimated from analysis of covariance (ANCOVA) model that included baseline score as a covariate.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug and had baseline, post-baseline ITSQ data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LY900014
Number analyzed (Participants) | 160
score on a scale | 16.9 (1.55)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 14 weeks)
Description: All participants who received at least one dose of study drug.
Arm/Group | LY900014
All-Cause Mortality (participants affected / at risk) | 0/176
Serious Adverse Events (participants affected / at risk) | 3/176
Other Adverse Events (participants affected / at risk) | 0/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=176)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04605991/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT04605991/SAP_001.pdf